CLINICAL TRIAL: NCT01207154
Title: BIS-guided Conscious Sedation for Awake Intubation
Brief Title: Feasibility of Using Depth-of-sedation Measuring Equipment (BIS) to Guide Awake Fibreoptic Intubation
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty in Recruitment due to lack of investigators and suitable patients
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 10/H0724/40
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2013-05

CONDITIONS: Known Difficult Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BIS guidance: Sedation guided according to a predetermined BIS level
- Clinical sign guided: Sedation guided by clinical signs

SUMMARY:
The purpose of this study is to determine whether or not a device which measures depth of anaesthesia and sedation can be used to assist in the sedation of patients who must have breathing tubes positioned in their airways before general anaesthesia

DETAILED DESCRIPTION:
As part of a general anaesthetic, patients frequently have a breathing tube positioned in their trachea (windpipe) and this is usually performed after they have gone to sleep. For some patients however, problems with their mouths or neck may mean it is safer for the tube to be placed before they are asleep and this is performed with the aid of sedation. The level of sedation is vital. Patients must be adequately sedated to tolerate instruments in their airway yet at the same time patients must not be oversedated so that they fall asleep or stop breathing. Assessments using clinical endpoints of sedation are subjective, vary between observers and patients and do not prevent episodes of undersedation or oversedation. An objective measure of sedation depth would facilitate safe awake intubation. Previous studies demonstrate that commercially available depth of anaesthesia monitors can be used to measure depth of sedation too. We wish to find out if one such monitor can be used to help achieve the right level of sedation in patients who must have an awake intubation as part of their anaesthetic. Depth of sedation guided awake intubation has not been described previously. The current study would comprise two parts. In the first, we will measure sedation depths correlating with clinical signs of optimal sedation using propofol and remifentanil in a cohort of patients requiring awake intubation. In the second part, we will titrate sedation in a cohort of patients requiring awake intubation to the 25th-75th centile of the values obtained in the first part and determine the adequacy of the conditions achieved. Patients who are likely to require an awake fibreoptic intubation will be identified when they attend for their preadmission assessment. Patients requiring certain surgical procedures, by their very nature, will have a high chance of being deemed to require an awake intubation on the day of admission. Such procedures, for example, include (but are not limited to) revision surgery for patients who have previously undergone Maxillofacial reconstructive surgery and cervical spine neurosurgery for unstable neck disease. These patients will be given written information explaining that should they go on to require an awake intubation, they may be invited to participate in the study. This written material will thus be available to potential study participants for a period of two to four weeks prior to their admission. On the day of admission, patients who the anaesthetist decides will require an awake intubation and who are suitable for inclusion in the study will be approached by one of the researchers who will offer them the opportunity to be enrolled in the study. Informed consent will be obtained after patients have had the opportunity to ask any questions about the study. Awake intubation is associated with specific advantages, disadvantages and risks. Both groups of patients however will receive the same awake intubation technique as those not participating in the study. The first part of the study involves only the application of noninvasive forehead electrodes over and above the treatment patients would receive whether a study participant or not. In the second part of the study, participants will be sedated initially by titration to BIS values of depth of sedation to evaluate the usefulness of this measurement. If at any time, the level of sedation in any patient in this second group is deemed clinically inappropriate, the situation will be modified according to clinical criteria. Since clinically guided sedation is the usual standard of care, we feel again that attachment of the BIS electrodes is the only difference from the usual treatment that participants will experience. The BIS depth of anaesthesia monitor is CE marked and has been used safely on 34 million patients worldwide. Reliance on BIS measured depth of anaesthesia to the exclusion of clinical signs is no guarantee of clinically appropriate anaesthesia and so the same caveat must be applied to it's use to monitor sedation. In this study, monitoring of and adjustment of sedation by clinical signs will apply at all times as would occur without BIS monitoring. There are no risks associated with the use of forehead electrodes per se. Information will be rendered unidentifiable by not recording any information on data collection sheets which may identify patients. Data will be recorded on a spreadsheet, entered on a computer and kept only by the principle investigators.The data forms will be kept in a locked cupboard. No identifiable patient information will be kept after completion of the project and no participants will be identifiable from the published results.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III Patients scheduled for elective surgery and likely to need general anaesthesia and an awake fibreoptic intubation.
* Male or female patients aged from 18 to 79 years old will be included.
* Patients must be willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Patients under 18
* pregnant women
* patients requiring emergency surgery
* Patients of ASA status IV and V
* Inability to communicate
* Allergy to any of the drugs used, in particular remifentanil and propofol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring elective maxillofacial, ENT or cervical spine neurosurgery who also require awake fibreoptic intubation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
To determine if bispectral index (BIS) can be used to guide conscious sedation for awake fibreoptic intubation | 30 minutes
  Sedation is increased in increments until the patient will tolerate the procedure and maintain their own airway and oxygenation throughout the procedure. In the second part, sedation, instead of being based on clinical signs, will be initially adjusted according to the BIS values derived from part one of the study. Upon reaching the level of sedation corresponding with the target BIS value, the Steward score will be assessed and the procedure will continue as above if the patient is deemed optimally sedated clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Mridula Rai, MBBS FRCA MD, Principal Investigator — Oxford University Hospitals NHS Trust; Kevin D Johnston, MBChB BSc FRCA, Principal Investigator — Oxford University Hospitals NHS Trust; K K Ramaswamy, MBBS FRCA, Principal Investigator — Oxford University Hospitals NHS Trust; Alexander Marfin, MD FRCA, Principal Investigator — Oxford University Hospitals NHS Trust; Mansukh T Popat, FRCA, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- The John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom